CLINICAL TRIAL: NCT01118884
Title: Sedative Effects of Oral Midazolam in Comparison Promethazine With Nitrous Oxide/Oxygen on Behavior Management of Uncooperative Children Receiving Dental Treatment
Brief Title: Effects of Oral Midazolam in Comparison Promethazine With Nitrous Oxide for Uncooperative Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Sedighe Mozafar, Shahid Beheshti University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 171598
Record Dates: First submitted 2010-04-26; First posted 2010-05-07 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-04

CONDITIONS: Conscious Sedation
Keywords: Midazolam; Nitrous oxide; Behaviour management
MeSH Terms: interventions — Promethazine; Diphenhydramine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sedation (Experimental): 20 healthy uncooperative children aged 36-96 months were examined in a cross-over study design , each patient served as his/her own control. Each patient was assigned randomly to received 1 of 2 drug regimens for initial sedation session and the other regimen administered at second session which was one week later.
  Interventions: Drug: Promethazine

INTERVENTIONS:
Drug: Promethazine — Syrup ,1 mg/kg, oral , 30 minutes before dental procedure , its duration is 4-6 hours
  Other Names: Phenergan; Prothiazine; Promethegan; Romergan

SUMMARY:
The purpose of this study is to compare the safety and efficacy of sedation using orally administered midazolam and promethazine with nitrous oxide/oxygen in uncooperative children receiving dental treatments.

DETAILED DESCRIPTION:
The effectiveness of oral midazolam in pediatric dentistry is controversial. Usefulness of midazolam alone is limited to short-duration procedures, and we are needed to identify safe oral conscious regiments which permit longer duration procedures in dental treatments especially in Pediatric dentistry.

Promethazine is a long-acting (4-12 hr) anti-histaminic, H1 antagonist drug which acts as a central nervous system depressant and showing itself to be a weak anxiolytic drug.

The hypothesis to be tested is whether promethazine would improve the patients behavior during dental procedures without affecting vital signs, thus enabling longer periods of moderate or conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients who are in ASA class 1 group
* Age of the patients must be between 36-96 months
* Uncooperative children who are in groups 1 or 2 according to Frankel's classification

Exclusion Criteria:

* Tonsil hypertrophy
* History of allergies
* Drooling or nocturnal snoring

Ages: 36 Months to 96 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Behavior change | during dental treatment which is 30 minutes after drug ingestion
  Behavior evaluation was based on a scale proposed by Houpt et al. which establishes the following scores : sleep, movement, crying , overall behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Sedighe Mozaffar, Principal Investigator — Postgraduate student of Shahid Beheshti Medicine University
Locations (1):
- Dental school of Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province, Iran